CLINICAL TRIAL: NCT06095791
Title: Identification of Immunomodulators Associated With Atrial Fibrillation Reporting: Analysis of the WHO Pharmacovigilance Database
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: CaenUH_JF_1
Record Dates: First submitted 2023-09-08; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2022-08

CONDITIONS: Atrial Fibrillation
Keywords: Immunomodulators; Pharmacovigilance; Atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Immunologic Factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Immunomodulators with FDA approval on the 1st January 2023. — Disproportionnality analysis studying the association between immunomodulators with FDA approval on the 1st January 2023 and atrial fibrillation in the World Health Organization pharmacovigilance database.

SUMMARY:
Atrial fibrillation is the most prevalent sustained arrhythmia worldwide with a great morbimortality. Some populations are more at risk to develop atrial fibrillation like patients suffering from inflammatory diseases or patients suffering from cancers. This is at least explained by the inflammatory environment related to these both conditions. Many experimental studies and clinical studies support the role of inflammation and immunity in atrial fibrillation genesis by modulating atrial action potential et by promoting fibrosis.

Immunomodulators are drugs used to stimulate or inhibit the immune system for two main indications : cancers and immune disorder diseases which both promote atrial fibrillation. Due to their interactions with inflammation and immunity, immunomodulatores may further promote the risk of atrial fibrillation, particularly in a population already at risk.

Based on the World Health Organization global database, the main objective of this study is to investigate the association between immunomodulators and the occurrence of atrial fibrillation reported in the database.

A disproportionality analysis will be performed. It will aim to assess whether immunomodulators are associated with a greater risk of atrial fibrillation.

Secondary objectives aim to describe the cases of atrial fibrillation among immunomodulators associated with atrial fibrillation in the main analysis, to describe coprescription among immunomodulators associated with atrial fibrillation in the main analysis, to analyse the role of immunomoduloators medical indication in the overrisk of atrial fibrillation, and to try to highlight some immune mechanisms promoting atrial fibrillation regarding the immunomodulators associated with atrial fibrillation in the main analysis.

ELIGIBILITY:
Inclusion Criteria:

* Case reported in the World Health Organization (WHO) database of individual safety case reports to 01/09/2022
* Patients treated with FDA approved immunomodulators (approval the 1st January 2023).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Every patients in the World Health Organization (WHO) database of individual safety case reports to 01/09/2022 included with at least one immunomodulator.
Sampling Method: Non-Probability Sample
Enrollment: 4000000 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Association between atrial fibrillation and immunomodulators | Case reported in the World Health Organization (WHO) of individual safety case reports to September 2022
  A disproportionality analysis is carried out in multivariate analysis taking into account cofounding factors (factors known to promote atrial fibrillation).

SECONDARY OUTCOMES:
Descriptive analysis of the atrial fibrillation cases with immunomodulators significantly associated with atrial fibrillation in the primary analysis | Case reported in the World Health Organization (WHO) of individual safety case reports to September 2022
  The investigators describe the profile of cases of atrial fibrillation among immunomodulators associated with atrial fibrillation in the main analysis. We particularly focused on factors known to promote atrial fibrillation.
Identification of molecular/cellular pathway through mechanism of action of immunomodulators associated with AF in the primary analysis. | Case reported in the World Health Organization (WHO) of individual safety case reports to September 2022
  The aim is to suggest a physiopathology model focused on the role of immune system in atrial fibrillation genesis by taking into account the state of knowledge and the mechanisms suggested by the immunomodulators associated with atrial fibrillation in the main analysis.
Exploratory analysis: association between immunomodulators medical indication and atrial fibrillation. | Case reported in the World Health Organization (WHO) of individual safety case reports to September 2022
Descriptive analysis of the coprescription between immunomodulators associated with atrial fibrillation in the main analysis. | Case reported in the World Health Organization (WHO) of individual safety case reports to September 2022

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandre Joachim, Caen, Basse Normandie, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Alexandre J, Salem JE, Moslehi J, Sassier M, Ropert C, Cautela J, Thuny F, Ederhy S, Cohen A, Damaj G, Vilque JP, Plane AF, Legallois D, Champ-Rigot L, Milliez P, Funck-Brentano C, Dolladille C. Identification of anticancer drugs associated with atrial fibrillation: analysis of the WHO pharmacovigilance database. Eur Heart J Cardiovasc Pharmacother. 2021 Jul 23;7(4):312-320. doi: 10.1093/ehjcvp/pvaa037. PMID 32353110
- [Result] Lazzerini PE, Capecchi PL, Laghi-Pasini F. Systemic inflammation and arrhythmic risk: lessons from rheumatoid arthritis. Eur Heart J. 2017 Jun 7;38(22):1717-1727. doi: 10.1093/eurheartj/ehw208. PMID 27252448
- [Result] Guo Y, Lip GY, Apostolakis S. Inflammation in atrial fibrillation. J Am Coll Cardiol. 2012 Dec 4;60(22):2263-70. doi: 10.1016/j.jacc.2012.04.063. PMID 23194937
- [Result] Lazzerini PE, Laghi-Pasini F, Acampa M, Srivastava U, Bertolozzi I, Giabbani B, Finizola F, Vanni F, Dokollari A, Natale M, Cevenini G, Selvi E, Migliacci N, Maccherini M, Boutjdir M, Capecchi PL. Systemic Inflammation Rapidly Induces Reversible Atrial Electrical Remodeling: The Role of Interleukin-6-Mediated Changes in Connexin Expression. J Am Heart Assoc. 2019 Aug 20;8(16):e011006. doi: 10.1161/JAHA.118.011006. Epub 2019 Aug 19. PMID 31423933